CLINICAL TRIAL: NCT06878612
Title: A Clinical Trial to Evaluate the Safety, Tolerability, and Preliminary Antitumor Activity of a Polyphenol Whole Tumor Cell Vaccine in Patients With Advanced Malignant Solid Tumors
Brief Title: a Polyphenol Whole Tumor Cell Vaccine in Patients With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xingchen Peng (Other)
Responsible Party: Sponsor-Investigator, Xingchen Peng, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2435
Record Dates: First submitted 2025-02-26; First posted 2025-03-17 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Polyphenols; Cancer Vaccine; Advanced Solid Tumor
Keywords: polyphenols; whole tumor cell vaccine; advanced solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polyphenol whole tumor cell vaccine (Experimental): In this study, a group of three patients were subjected to a "3+3" dose climb, sequentially testing doses of 5×10*6, 2×10*7, and 5×10*7 cells/dose, with close monitoring of the patients during the climb and assessment of the occurrence of DLT events during the dose-limiting toxicity (DLT) cycle, and obtaining the previous group's safety data after evaluated before enrollment in the next dose group was initiated.
  Interventions: Biological: Polyphenol whole tumor cell vaccine

INTERVENTIONS:
Biological: Polyphenol whole tumor cell vaccine — 3 patients enrolled in each dose group, and planned dose groups of 5 x 10*6, 2 x 10*7, and 5 x 10*7 cells/dose. The dosing regimen consisted of 5 doses of basal immunization and subsequent individualized treatment. In the basal immunization, the administration times were D0, D14, D28, D42, and D56. After completion of the 5 doses of basal immunization, the subsequent individualized treatment was decided by the investigator based on the subject's tumor assessment, i.e., 1 vaccination per month for a total of 4 doses.

SUMMARY:
This project intends to carry out phase I clinical studies on the basis of the previous work, initially exploring the possible effective dose, evaluating its safety and tolerability, with a view to achieving long-term control of the disease, which is expected to provide more options for the treatment of patients with advanced malignant solid tumors. The development of this project will provide new ideas, strategies and theoretical basis for the research and development of whole tumor cell vaccines; at the same time, it is expected to obtain original new drugs with independent intellectual property rights.

DETAILED DESCRIPTION:
Malignant solid tumors are malignant tumors that originate in epithelial tissue (carcinoma), mesenchymal tissue (sarcoma), or the nervous system (glioma, etc.). According to Global Cancer Statistics 2022, there will be 19.96 million new cancer cases and 9.74 million new deaths globally in 2022, with solid tumors accounting for the majority of these cases. Overall, the annual global cancer incidence rate continues to trend upward, and the number of new cancers in 2050 is expected to increase to 35.3 million cases. Cancer remains a major health challenge globally, with serious implications for human life safety and quality of life.

Tumor vaccines are a promising immunotherapeutic modality to achieve inhibition of tumor growth and metastasis by utilizing the body's immune system to trigger a specific anti-tumor immune response. In recent years, impressive progress has been made in the development of tumor vaccines, and hundreds of such vaccines are currently under development and in clinical trials. These vaccine types are mainly tumor cell vaccines, dendritic cell vaccines, peptide vaccines, oncolytic viral or bacterial vector vaccines, and nucleic acid vaccines. Typically, the effectiveness of tumor vaccines relies on the availability of a sufficiently large number of tumor antigens to stimulate the innate immune system, and the ability to achieve antigen cross-presentation and T-cell immune activation. However, most tumor vaccines developed at this stage do not contain complete antigenic information, which affects the clinical efficacy of the vaccine and hinders application expansion. In order to avoid the problem of immune escape caused by insufficient immune stimulation due to the lack of a sufficient number of tumor antigens, the development of autologous tumor cells and the retention of complete specific tumor-associated antigens have become the key to the development of personalized vaccines.

Whole tumor cell vaccine (TCV) is a classic individualized tumor immunotherapy, and its advantage lies in the inclusion of the patient's own full series of tumor-associated antigens, which can simultaneously target multiple unknown and known tumor antigens optimally, thus avoiding immune escape caused by the loss of tumor antigens, and has an important application prospect for the inhibition of tumor development, progression and recurrence. It has important application prospects for inhibiting tumor occurrence, development and recurrence. Its mechanism of action is to introduce tumor antigens into the patient's body in order to overcome tumor-induced immunosuppression, enhance immunogenicity, activate the patient's own immune system, induce the body's cellular and humoral immune responses, and achieve the goal of controlling or clearing the tumor. Although these strategies are promising, it is still difficult to retain intact tumor antigens and effectively trigger anti-tumor immune responses during vaccine preparation. In addition, since vaccines made from intact tumor cells usually fail to elicit an effective immune response, in order to improve their immunogenicity as vaccines, scientists have been exploring adjuvant-related approaches to introduce various interventions to enhance their immune potential. However, these methods are usually complex and time-consuming, and therefore, there is an urgent need to develop new concepts and technologies through interdisciplinary intersections to achieve on-demand immunopotentiation of TCVs.

Recently, the team of investigators developed a novel strategy of encapsulating tumor cells by metallic polyphenol nanocoatings and further constructed a whole-cell vaccine (referred to as LMP vaccine) using bacterial lipopolysaccharide (LPS) with surface modification as a vaccine adjuvant. In this study, by constructing a single-cell coating of plant polyphenols, all neoplastic antigens of the encapsulated tumor cells were preserved, and upon uptake by dendritic cells, the LMP vaccine released manganese ions and tumor antigen components inside the dendritic cells to stimulate the innate immune pathway STING, which synergistically with the tumor antigens facilitated the maturation of the dendritic cells and further presented the tumor antigen signals to the T cells, resulting in an enhanced The research results of LMP vaccine were published in Angewandte Chemie International Edition in 2024 and selected as "Hot Paper", which gained wide attention. The study used C57BL/6 mice to establish a B16F10 melanoma model, and after inoculation with tumor cells on day 0, the mice were injected subcutaneously with the LMP vaccine on days 3, 6, 9, and 15. The results showed that tumor growth was significantly inhibited in the LMP vaccine group compared with the PBS control group, and the average tumor volume was only 350 mm³ on day 20, while the average tumor volume of the PBS group was more than 1,200 mm³. The mean tumor volume of the PBS group exceeded 1200 mm³. In addition, when the LMP vaccine was combined with anti-programmed cell death ligand 1 (anti-PD-L1), the therapeutic effect was even more pronounced, and the tumor volume of all mice receiving the combined treatment was significantly reduced, with the mean tumor volume reduced to less than 100 mm³, demonstrating a synergistic tumor-suppressive effect. In addition, the investigators paid special attention to the safety of the LMP vaccine, especially the inactivation of tumor cells and the risk of secondary tumorigenesis. The results showed that the LMP vaccine was successfully inactivated by encapsulation of metal polyphenol nanocoatings during the preparation of tumor cells, which lost their proliferation ability after injection. Through in vivo observations in mice for up to 27 days, the investigators found that mice receiving the LMP vaccine did not show any signs of tumor growth, whereas mice in the control group rapidly developed significant tumors, with tumor volumes exceeding 1,400 mm³ within 27 days. In addition, by histopathological analysis of major organs (heart, liver, spleen, and kidneys), H&E staining showed no significant differences in organ histology between the different treatment groups of mice, suggesting that the LMP vaccine did not cause significant tissue damage. Key blood biochemical analyses, including aspartate aminotransferase (AST), alanine aminotransferase (ALT), albumin (ALB), creatine kinase (CK), creatinine (CREA), and urea (UREA), were all within the normal reference ranges, which further confirmed the systemic safety of the LMP vaccine. Together, these data indicate that the LMP vaccine provides an effective anti-tumor immune response as well as good biocompatibility and safety, does not cause secondary tumorigenesis, and provides a solid safety foundation for clinical application. In summary, the results show that LMP vaccine is biosafe and can inhibit primary tumor growth and metastasis. In combination with anti-programmed cell death ligand 1 (anti-PD-L1), it showed synergistic tumor inhibition effects, which is important for achieving superior anti-tumor therapeutic effects in the clinic.

This project intends to carry out phase I clinical studies on the basis of the previous work, initially exploring the possible effective dose, evaluating its safety and tolerability, with a view to achieving long-term control of the disease, which is expected to provide more options for the treatment of patients with advanced malignant solid tumors. The development of this project will provide new ideas, strategies and theoretical basis for the research and development of whole tumor cell vaccines; at the same time, it is expected to obtain original new drugs with independent intellectual property rights.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 years (including borderline values) at screening.
2. Advanced metastatic malignant solid tumors (skin or limb melanoma/head and neck tumors/soft tissue tumors, etc.) confirmed histologically or cytologically, with previous failure of second-line or higher treatment (refer to the China Clinical Oncology (CSCO) Melanoma Guidelines 2024, CSCO Head and Neck Tumor Guidelines 2024, and CSCO Bone and Soft Tissue Tumor Guidelines.

   Note: ① Advanced metastatic melanoma: first-line standard treatment includes dacarbazine/timozolomide ± platinum ± endo, and dabrafenib + trametinib is recommended if the BRAF V600 mutation is carried. Second-line treatment may be considered with a different drug therapy than first-line treatment, and if PD-1 monoclonal antibody is not used in the first line, pabolizumab or treprotilizumab is recommended in the second line. If tumor reduction is urgently needed, targeted drugs or chemotherapy combination regimens (paclitaxel/albumin paclitaxel ± platinum ± antivascular drugs) are preferred in the second line. If NRAS mutation is carried, tulolametinib (HL085) is recommended.

   (ii) Advanced metastatic head and neck tumors: first-line standard treatment includes pembrolizumab + cisplatin/carboplatin + 5-Fu, pembrolizumab (CPS ≥ 1), cisplatin/carboplatin + 5-Fu + cetuximab, cisplatin + docetaxel + cetuximab, and cisplatin/carboplatin + paclitaxel ± cetuximab. Second-line or salvage therapy is recommended, such as nabulizumab.

   (iii) Advanced metastatic soft tissue sarcoma: first-line standard treatment includes doxorubicin ± isocyclophosphamide chemotherapy, and second-line treatment is based on the specific type of chemotherapy or amilorotinib targeted therapy.
3. Presence of at least 1 measurable or evaluable lesion according to RECIST v1.1 criteria.
4. Eastern Cooperative Oncology Group (ECOG) physical status score: 0 to 2.
5. Expected survival ≥ 3 months.
6. Good function of major organs, and the following requirements are met by the examination indexes within 7 days prior to receiving treatment:

   ① Hemoglobin ≥80 g/L; neutrophil count >1.5×109/L; platelet count ≥80×109/L;

   ② Total bilirubin ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 × ULN; if there are liver metastases, ALT or AST ≤ 5 × ULN;

   ③ Creatinine (SCr) ≤ 1.5 × ULN or creatinine clearance (CRCI) ≥ 60 mL/min (Cockcroft-Gault formula) (see 16.6 Appendix VI);

   ④ Prothrombin time (PT), International Normalized Ratio (INR) ≤ 1.5 x ULN (unless warfarin anticoagulation is being used).

   ⑤ Cardiac function: left ventricular ejection fraction (LVEF) ≥50%.
7. Able to understand and voluntarily sign a written informed consent before the trial.

Exclusion Criteria:

1. Patients with a prior history of other tumors, except for cured and non-recurrent basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, cervical cancer in situ, gastrointestinal intramucosal carcinoma, and other histories of malignancies deemed by the investigator to be eligible for enrollment.
2. Patients with known concomitant cardiac clinical conditions or diseases that are not well controlled, e.g., New York Heart Association (NYHA) class II or higher heart failure (see 16.5 Appendix V), unstable angina, myocardial infarction within 6 months, supraventricular or ventricular arrhythmias that are clinically significant and require treatment or intervention.
3. Patients with previous and current objective evidence of asthma, history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, and severely impaired lung function.
4. Have any uncontrollable clinical disease (e.g., respiratory, circulatory, digestive, neurologic, hematologic, genitourinary, endocrine system disorders) or psychiatric disease (e.g., depression, schizophrenia) or other significant illnesses assessed by the investigator as preventing the provision of informed consent, interfering with the interpretation of the trial results, potentially posing a risk to subjects by participating in this trial, or otherwise otherwise interfere with achieving the purpose of the study.
5. Have any active autoimmune disease or a history of autoimmune disease including, but not limited to, immune-related neurological disorders, multiple sclerosis, autoimmune (demyelinating) neuropathies, Guillain-Barre Syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease including Crohn's disease and ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis-relaxation (TEN) or Stevens-Johnson syndrome (except for type I diabetes on stable doses of insulin).
6. Allergy to the test drug (including any excipients). Prior history of severe allergy to any drug, food, or vaccination, such as anaphylaxis, anaphylactic laryngeal edema, anaphylactic dyspnea, anaphylactic purpura, thrombocytopenic purpura, and localized anaphylactic necrotic reaction (Arthus reaction).
7. the existence of intradermal injection contraindications: ① injection site inflammation, trauma ulceration. ② severe bleeding, coagulation tendency, platelets or coagulation factors significantly reduced. ③ Any abnormalities or permanent body art (e.g., tattoos) at the vaccination site that, in the opinion of the investigator, would prevent observation of local reactions at the vaccination site.
8. Participation in other drug or device clinical trials within 3 months prior to screening.
9. Major surgery (minor surgery such as catheterization, protocol-required biopsy procedures, etc. is not an exclusion criterion) within 4 weeks prior to the first dose of vaccination or less than 14 days of elimination of the effects of surgery or trauma prior to enrollment, radiotherapy, targeted, immune checkpoint inhibitors, interferon, live/live attenuated vaccines, and other treatments.
10. Patients who have not recovered to NCI CTCAE ≤ grade 1 for antitumor therapy-related adverse reactions (except alopecia) after previous antitumor therapy.
11. Subjects on systemic therapy with corticosteroids (>10 mg/day of prednisone or equivalent dose of other glucocorticoids) or other immunosuppressive agents within 14 days prior to the first dose of vaccination. Inhaled or topical steroids and adrenal hormone replacement at doses ≤ 10 mg/day prednisone efficacy dose are allowed in the absence of active autoimmune disease.
12. Known hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), and syphilis infections, or positive hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus antibody (HCVAb), HIV antibody, and syphilitic spirochete (TP) antibody test at screening: HBsAg (+) or HBcAb (+), and HBV DNA copy number ≥ 2000 IU/mL (or the lower limit of positive test values at the host research center); HCVAb positive and HCV RNA ≥ ULN at the host research center.
13. Patient has a history of active tuberculosis (TB) (patients suspected of having active TB need to be examined on chest X-ray, sputum, and excluded by clinical signs and symptoms) or active TB; or severe acute or chronic infection requiring systemic therapy.
14. History of substance abuse or known medical, psychological, or social conditions such as alcohol or drug abuse.
15. Pregnant or breastfeeding women with a screening period up to 12 months after the full course of drug injection, a planned pregnancy in a female subject or a planned pregnancy in the partner of a male subject.
16. Any other factors that, in the opinion of the investigator, make it inappropriate for the subject to enter this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability. | From the time of the first dose to 14 days after the last vaccination.
  DLT was defined as a therapeutic drug-related TEAE or clinically significant abnormal laboratory test occurring during the DLT observation period as follows:1) Hematologic toxicity:① ≥ grade 4 neutropenia lasting more than 5 days (after symptomatic treatment);② ≥ grade 3 febrile neutropenia;③ ≥ grade 4 thrombocytopenia;④ ≥ grade 3 thrombocytopenia with bleeding tendency;⑤ ≥ grade 4 anemia.2) Non-hematological toxicity:① ≥ grade 3 non-hematologic toxicity shall be considered DLT, except for the following:a) Alopecia of any grade;b) Grade 3 nausea, vomiting, or diarrhea, if well controlled within 72 hours;c) Grade 3 fatigue < 7 days;d) Abnormal laboratory tests without clinically relevant signs or symptoms.② Any concurrent grade ≥2 total bilirubin elevation and grade ≥3 alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation (Hay's rule); for patients with liver metastases, an AST or ALT > 8 x upper limit of normal (ULN); and an AST or ALT > 5 x ULN for ≥14 days.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | From the time when the patients were enrolled in the study to the whole study completion, an average of 1 year.
  It refers to the proportion of patients whose tumors have shrunk to a certain extent and remained so for a certain period of time. It is a direct indicator to measure the anti-tumor activity of drugs.It is usually calculated as the percentage of the sum of the number of patients with complete response (CR) and partial response (PR) in the total number of patients.
Progression-free survival (PFS). | From the time when the patients were enrolled in the study to the whole study completion, an average of 1 year.
  PFS was defined as the time interval from the initiation of study treatment to the first occurrence of PD or death due to any cause.
Overall survival (OS). | From the time when the patients were enrolled in the study to the whole study completion, an average of 1 year.
  OS was defined as the time interval from the start of study treatment to the death of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Professor, Principal Investigator — Department of Biotherapy, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan Universit, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No